CLINICAL TRIAL: NCT01586741
Title: A Prospective Randomized Study to Evaluate Two Different Surgical Methods for Treatment for Abdominal Wall Diastasis
Brief Title: A Study to Evaluate Two Different Surgical Methods for Treatment for Abdominal Wall Diastasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Peter Emanuelsson, MD, consultant in plastic surgery, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009/227-31/3/PE/96
Record Dates: First submitted 2011-11-21; First posted 2012-04-27 (Estimated); Results first posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-11

CONDITIONS: Abdominal Hernias and Other Abdominal Wall Conditions; Post-operative Pain; Recurrence
MeSH Terms: conditions — Hernia, Abdominal; Pain, Postoperative; Recurrence | interventions — Wound Healing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Polypropylene mesh (Active Comparator): Reconstruction of the abdominal wall diastasis with insertion of a polypropylene mesh on 30 patients.
  Interventions: Procedure: Quill suture application for repair or polypropylene mesh
- quill suture (Active Comparator): Reconstruction of the abdominal wall diastasis with double row absorbable suture ( Quill Self-retaining system) on 30 patients.
  Interventions: Procedure: Quill suture application for repair or polypropylene mesh
- conservative treatment (No Intervention): Regular abdominal exercises workout for three months for 30 patients.

INTERVENTIONS:
Procedure: Quill suture application for repair or polypropylene mesh — The first arm may be insertion of the-mesh The second arm may double row- suture The third arm may be conservative -training
  Other Names: Quill suture; And Soft mesh Polypropylene mesh
  Arms: Polypropylene mesh; quill suture

SUMMARY:
This is a three armed prospective randomized trial that will compare two different surgical techniques for reconstruction of the abdominal wall diastasis with a conservative treatment procedure.

The study hypothesis:

Which surgical approach provides the safest and best long term results for patients with abdominal wall diastasis either the insertion of net alternative with a double row suture or exercise alone?

DETAILED DESCRIPTION:
The conservative control group will receive a special training program for abdominal muscle training for 3 months,and all groups wearing girdle for 3 months.

All patients examined with a CT scan before randomization and then a Biodex measurement of abdominal muscle strength.

All patients must also complete the SF-36 (scientifically tested instruments to measure self-reported physical and mental health) and VHPQ (ventral hernia Pain Questionnaire).

Two-thirds of patients receive surgery and followed up with a 3 month and 1-year control.At 1 year of control, all go through a CT scan and a Biodex measurement of muscle strength.

The control group followed up after one and half months and 3 months. In the surgery group, patients may not know what reconstruction they received before the final assessment after 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Abdominal wall diastasis> 3 cm
2. Discomfort or tenderness in the abdominal wall
3. Desire for abdominal wall reconstruction
4. Women have undergone at least one birth
5. Smoking cessation 1 month pre-and 3 months post-operatively

Exclusion Criteria:

1. <18 years old
2. Ongoing pregnancy
3. Ongoing breastfeeding
4. Current immunosuppressive therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulf S Gunnarsson, professor, Study Director — Karolinska Institutet
Locations (1):
- Clintec, Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Derived] Emanuelsson P, Gunnarsson U, Strigard K, Stark B. Early complications, pain, and quality of life after reconstructive surgery for abdominal rectus muscle diastasis: a 3-month follow-up. J Plast Reconstr Aesthet Surg. 2014 Aug;67(8):1082-8. doi: 10.1016/j.bjps.2014.04.015. Epub 2014 May 2. PMID 24880577

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Quill Suture | Polypropylene Mesh | Conservative Treatment
Started | 28 | 29 | 32
Completed | 27 | 29 | 30
Not Completed | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polypropylene Mesh | Quill Suture | Conservative Treatment | Total
Number analyzed (Participants) | 29 | 28 | 32 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 28 | 31 | 88
  >=65 years | 0 | 0 | 1 | 1
Age, Continuous [Median (Full Range); unit: years] | 42 [27 to 62] | 39.6 [24 to 61] | 44.2 [28.9 to 66.9] | 41.9 [24 to 66.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 32 | 87
  Male | 1 | 1 | 0 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 29 | 28 | 32 | 89

OUTCOME MEASURES:

1. Primary Outcome: Recurrence of Diastasis One Year Post-operatively That Indicated by CT Scan or Clinical Investigation.
Description: All patients go through a CT scan and clinical examination one year after surgery
Time Frame: follow-up 1 year after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Polypropylene Mesh | Quill Suture | Conservative Treatment
Number analyzed (Participants) | 29 | 27 | 30
Participants | 2 | 3 | 26

2. Secondary Outcome: Adverse Event Indicated in Case Report Formulary During the First 12 Months
Description: adverse event categorize as superficial wound infection, seroma, fistula or deep wound infection
Time Frame: follow-up 1 year after surgery
Reporting Status: Not Posted, anticipated posting 2020-11

3. Secondary Outcome: Pain Post Operatively Measured by the VHPQ Questionnaires
Description: The validity and reliability of the VHPQ make it a useful tool in assessing postoperative pain and patient satisfaction.
  PMID:
  22446989 PubMed - as supplied by publisher
Time Frame: follow-up 1 year after surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Quill Suture | Polypropylene Mesh | Conservative Treatment
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/27 | 0/29 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes